CLINICAL TRIAL: NCT03435354
Title: Impacting Child Physical and Mental Health Outcomes in Congenital Heart Disease: A Randomized, Controlled Trial of Enhanced Physical Activity Support in Clinical Care
Brief Title: Enhanced Physical Activity Support in Congenital Heart Disease Clinical Care
Acronym: PAToolKit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Stollery Children's Hospital (Other); London Health Sciences Centre (Other); CHEO Family Forum (Unknown); Canadian Congenital Heart Alliance (Other); Ontario Child Health Support Unit (Unknown)
Responsible Party: Principal Investigator, Dr. Pat Longmuir, Scientist, Assistant Professor, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17/191X
Record Dates: First submitted 2018-01-31; First posted 2018-02-19 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Congenital Heart Disease
Keywords: Physical activity; Quality of life; Activity motivation; Children; Adolescents; Cluster-randomized trial
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster-randomized trial, with randomization by within each site by week (i.e., site-week)
Who Masked: Outcomes Assessor
Masking Description: Those conducting the post-intervention assessments will be blind to study group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Physical activity counselling during cardiac clinic visit with additional supports for community physical activity and access to a kinesiologist.
  Interventions: Behavioral: Physical activity counselling
- Usual Care (No Intervention): Cardiac clinic visit with usual care but no physical activity counselling

INTERVENTIONS:
Behavioral: Physical activity counselling — Clinician counselling about physical activity using standardized tools to promote daily physical activity.
  Other Names: PA counselling
  Arms: Intervention

SUMMARY:
Our cluster randomized controlled trial of a novel clinical practice change will IMPACT the physical activity (PA) of children living with congenital heart defects (CHD) through our

Innovative and pragmatic approach to systematically incorporate PA counselling within each clinic visit. Long-term, the focus is to prevent or treat the most common secondary morbidities of these patients (atherosclerosis, anxiety, depression) through enhanced PA. We have previously shown that home-based, PA interventions can increase daily PA and enhance PA motivation, motor skill and fitness when delivered via an intensive research intervention. Our objectives for this study are to

Measure the feasibility and efficacy of PA counselling using clinical resources among paediatric CHD patients (daily PA, PA motivation, competence, quality of life) and on clinic systems (% patients counselled, clinic/kinesiology personnel support required, clinic visit time, # of PA questions). Our

Patient-empowering, ready-to-use, self-explanatory "tool kit" of clinician PA resources and patient/family/clinician friendly searchable electronic PA database will be used to promote the

Active lifestyles that are critically important to physical/mental health, peer socialization & childhood growth/development. 90% of children are not active enough for optimal health.

We initially target children with CHD because they are less active than peers, and their most important secondary morbidities can be prevented or treated through PA. Our

Collaborative approach with patients, their families and leaders in paediatric cardiac healthcare will optimize our "PA tool kit" and novel practice change for

Translation to all paediatric CHD healthcare systems (primary, secondary, tertiary) through our pan-Canadian Cardiac Kids Quality of LIFFE Research and Knowledge Exchange Network, a collaborative of 10 patient/family support networks and 10 paediatric cardiac clinics in 6 provinces focused on Learning, Independence, Friends, Fitness & Emotional health (LIFFE).

DETAILED DESCRIPTION:
Inactive lifestyles have a huge cost to Canadians' health, our economy and healthcare system (3.7% of total healthcare costs, 2009=$6.8B19). If 10% of Canadians were more active, 25-yr healthcare costs would drop by $2.6B, $7.5B would be added to our economy, & 550,000 fewer Canadians would live with chronic disease. Congenital heart disease (CHD) is the most common congenital condition (12/1000 births) and a major health burden. 90% of CHD children live 4 to 8 decades with a 3-5X higher risk for atherosclerosis, anxiety or depression. Physical activity is known to decrease these important health risks. <10% of Canadian children are active enough for optimal health and, regardless of severity, CHD children are even less active. Individualized kinesiology support can improve physical activity (PA) skill, confidence and participation among CHD children but exceeds current clinical care resources. In response, our team of patients, parents, and clinicians developed a "tool kit" of 12 child/family-friendly PA resources to enable clinicians to better address the most important PA issues for these patients. Our randomized, controlled trial will evaluate a clinical practice change (systematic PA counselling with the PA tool kit plus PA in CHD database) on patient PA and health system outcomes in small (London), medium (Ottawa) and large (Edmonton) paediatric cardiac clinics. Randomization will be by week within each study site to prevent potential intervention cross contamination between children in clinic at the same time. Primary outcome is daily pedometer steps over 1 week. Secondary outcomes are quality of life (PedsQL), physical literacy (CAPL screen) and PA motivation (CSAPPA). Health system outcomes will be: % patients receiving intervention, clinic visit time, # of non-clinic contacts about PA, and need for kinesiology referral. Patient outcomes will be assessed during the CHD clinic visit and at 6 months, with pedometer steps also measured each month. We will enroll consecutive CHD patients with moderate or severe CHD, 5 - 17 yrs, & no other diagnosis affecting PA. Based on our data from previous PA studies among CHD patients and anticipating 10 patients/month, we would require 15 months of data collection (10% dropout) to obtain the 136 complete data sets required to provide 80% power to detect a clinically meaningful increase in daily PA of 1000 steps/day. Repeated measures ANOVA will evaluate study group impact (control/intervention) on pedometer steps. Secondary ANCOVA models will adjust for age, sex, treatment history and clinic site (Ottawa, London, Edmonton).

Our research team combines expertise in clinical intervention trials (Longmuir) and study design and analyses (Willan) with patient (Graham) & family (Rouble) experience plus > 60 years of clinical expertise (Lougheed, Norozi, Mackie). All investigators have previous experience leading multi-site research projects and supervising graduate students. Graham (Can. Congenital Heart Alliance) will ensure intervention relevance and scalability to all Canadian CHD patients. CHEO Family Forum (Rouble) will provide parent input. Through this study, we will advance knowledge of healthy, active lifestyles & PA support for CHD patients & the health system impacts of current practice recommendations to promote PA to CHD patients at every clinical encounter.

ELIGIBILITY:
Inclusion Criteria:

* All patients 5 to 17 years with CHD diagnoses classified as moderate or severe in complexity by the American College of Cardiology / American Heart Association joint guidelines.

Exclusion Criteria:

* Cardiac intervention (catheterization or surgery) in preceding 6 months. Syndrome/diagnosis affecting physical activity (e.g., developmental disability) or the ability to complete the assessment questionnaires.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in daily physical activity | Baseline then first week of each month for 6 months
  Pedometer step counts per day

SECONDARY OUTCOMES:
Change in physical activity adequacy and predilection | Baseline, 6 months
  Children's Self-Perceived Adequacy and Predilection for Physical Activity Scale (total score, range 20 to 80 points, higher values are a better outcome).
Change in quality of life | Baseline, 6 months
  Pediatric Quality of Life Inventory (PedsQL), score range 0 to 100, higher score is better quality of life
Change in physical literacy | Baseline, 6 months
  PLAY Tools Run2 and screening question

OTHER OUTCOMES:
Clinic visit time | Baseline
  Time from arrival to departure of patient for clinic visit
Number of PA encounters | Through study completion on average 6 months
  Number of times that patients contact the clinic between clinics for reasons related to physical activity
Delivery of PA counselling | Through study completion, on average 6 months
  Proportion of intervention patients who receive enhanced physical activity counselling during clinic visit
Advanced PA counselling | Through study completion, on average 6 months
  Proportion of intervention patients who are referred to kinesiologist for additional support

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Longmuir, PhD, Principal Investigator — Scientist
Locations (3):
- Canada (3):
  - Stollery Children's Hospital, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Study is funded by CIHR. Data is required to be shared upon completion of the project.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Longmuir PE, Lougheed J, Mackie AS, Norozi K, Yaraskavitch J, Chappell A, Dempsey A, Blais A, Foshaug R, Willan A, Graham J. In-Clinic Activity Promotion for Children With Congenital Heart Disease: Randomized Clinical Trial. CJC Pediatr Congenit Heart Dis. 2025 Feb 5;4(3):150-159. doi: 10.1016/j.cjcpc.2025.01.003. eCollection 2025 Jun. PMID 40933783